CLINICAL TRIAL: NCT04162483
Title: Safety and Performance of the Neuroform Atlas™ Stent System in Patients Requiring Stent Assisted Intracranial Aneurysm Treatment in France - A National, Retrospective Multi-center Registry
Brief Title: Safety and Performance of the Neuroform Atlas™ Stent System
Acronym: ATLAS-FR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: T4062
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Neuroform Atlas Stent System — Stenting Assisted coiling procedure

SUMMARY:
The objective of this retrospective study is to describe in real-life settings the clinical practice, utilization and the treated population outcomes at 1-year (12-16 months) follow-up at selected, representative centers in France.

DETAILED DESCRIPTION:
This proposed ATLAS FR study will be a retrospective review conducted to expand our knowledge of the clinical outcomes in subjects treated in France between 01 February 2017 and 01 March 2018.

This will provide a comprehensive data set that is specifically representative of the Atlas stent use in France.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had undergone a stent assisted intracranial aneurysm coiling with Neuroform Atlas for the treatment of intracranial aneurysm(s) between 1st Feb 2017 and 1st March 2 018.
* Patient and/or their representative have/has received the written information concerning the study and not expressed opposition to the collection of his data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects treated in one of the French Sites participating to the registry and who have been treated with Neuroform Atlas for the treatment of intracranial aneurysm(s) between 01 February 2017 and 01 March 2018.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
permanent morbidity and mortality rate | up to 12-16 months post-procedure
  any major ipsilateral stroke or neurological death

SECONDARY OUTCOMES:
AEs and device malfunctions | peri-procedure
  All intra-procedural AEs and device malfunctions
Efficacy Endpoint with mRS | immediately post-procedure and at 12-16 months post procedure
  Proportion of aneurysms with Raymond-Roy Occlusion Class I, II or III
Retreatment | up to 12-16 months
  Occurence of re-treatment
Subarachnoid hemorrhage (SAH) | Up to 12-16 months
  Occurence of SAH
Aneurysm rupture/re-rupture | Up to 12-16 months
  Occurence of Aneurysm rupture/re-rupture
SAEs resulting in neurological death | Up to 12-16 months
  Rate of SAEs resulting in neurological death
device-related SAEs | Up to 12-16 months
  Occurence of device-related SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Houdart, MD, Principal Investigator — Hopital Lariboisière
Locations (1):
- CHU Gui de Chauliac, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided